CLINICAL TRIAL: NCT05768607
Title: Evaluation of the Results of Laparoscopic Extraperitoneal ( Modified) Burch
Brief Title: Laparoscopic Extraperitoneal ( Modified) Burch Colposuspension
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Principal Investigator, Süleyman Salman, Associate Professor, Gaziosmanpasa Research and Education Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GaziosmanpasaTREHz
Record Dates: First submitted 2023-01-27; First posted 2023-03-14 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Stress Incontinence, Female
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Intervention Model Description: Normally patients with stress urinary incontinence undergoes laparoscopic burch operation if transvaginal sling surgery was not planned. Here in our study group the assigned surgery type applied to study group is extraperitoneal ( modified) burch operation which is performed by not interfering with the abdominal cavity. By the way our study is an interventional study and it is planned to discuss both the anatomic and functional results of this technique.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients undergone Laparoscopic Extraperitoneal Burch Colposuspension (Other)
  Interventions: Procedure: Quality of Life QUESTIONNAIRE (SF36); Procedure: INCONTINENCE IMPACT QUESTIONNAIRE (IIQ-7); Procedure: UROGENITAL DISTRESS INVENTORY (UDI - 6)

INTERVENTIONS:
Procedure: Quality of Life QUESTIONNAIRE (SF36) — Units of a scale of the patients will be compared pre and postoperatively by using SF36
Procedure: INCONTINENCE IMPACT QUESTIONNAIRE (IIQ-7) — Units of a scale of the patients will be compared pre and postoperatively by using IIQ-7
Procedure: UROGENITAL DISTRESS INVENTORY (UDI - 6) — Units of a scale of the patients will be compared pre and postoperatively by using UDI - 6

SUMMARY:
Urinary incontinence is a very common problem in women and can be seen at any age. Laparoscopic burch operation has been shown to be an effective, convenient and safe method in women with stress incontinence. Laparoscopic Burch operation is less invasive because it is advantageous in terms of hospitalization time, blood loss, pain and recovery time, but the disadvantage is the procedure time. Modified extraperitoneal technique may be a good method for lowering the procedure time.

DETAILED DESCRIPTION:
In the research; The pre- and postoperative urodynamics of patients who underwent laparoscopic extraperitoneal (modified) burch operation in the Gynecology and Obstetrics Clinic of Istanbul Health Sciences University Gaziosmanpasa Training and Research Hospital will be compared. Surgical outcomes together with complications will also be assessed.

In addition, the QUALITY OF LIFE (SF36), which determines the quality of life of the patients related to the urinary system functions, and the UROGENITAL DISTRESS INVENTORY (UDI - 6), INCONTINENCE IMPACT QUESTIONNAIRE (IIQ-7) questionnaires that determine the effects of urinary incontinence, will be assessed preoperatively and postoperative 6 months of the patients.

ELIGIBILITY:
Inclusion Criteria:

* having stress urinary incontinence

Exclusion Criteria:

* having any kind of urogynecological surgery history
* having pelvic mass
* having endometrial or myometrial pathology
* having uterine prolapsus grater than grade 2
* benign obese

Ages: 25 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-01-17 (Actual); Primary Completion 2023-07-17 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
Surgical outcomes | 1 year
  Operation time in minutes
Surgical outcomes | 1 year
  Bleeding volume in milliliter
Preoperative and postoperative urodynamic result | 1 year
  First sensation of fluid filled in bladder in milliliter will be compared.
Preoperative and postoperative urodynamic result | 1 year
  First urge sensation due to fluid filled in bladder in milliliter will be compared.
Preoperative and postoperative urodynamic result | 1 year
  Maximum cystometric capacity in milliliter will be compared.
Preoperative and postoperative urodynamic result | 1 year
  Compliance in milliliter/cmH2O will be compared.
Preoperative and postoperative urodynamic result | 1 year
  Q max in milliliter/second will be compared.
Preoperative and postoperative urodynamic result | 1 year
  Voided volume of the patients in milliliter will be compared.
Preoperative and postoperative Quality of life Questionnaire | 1 year
  The domains assessed were pain, diet, speech, recreation, anxiety, mood, and overall QoL. Patients were asked to choose a Likert scale response (for example, 1 = no pain to 5 = severe pain) to a question on each domain and higher score represents better health. overall score ranges from 6 to 30. Pre and postoperative values will be compared.
Preoperative and postoperative UROGENITAL DISTRESS INVENTORY | 1 year
  Score ranges from zero to 18 and higher scores indicate more severe symptoms and INCONTINENCE IMPACT QUESTIONNAIRE (IIQ-7) in which SCORES RANGES FROM 0 TO 21 AND a higher score indicates more severe symptoms and lower quality of life. Pre and postoperative values will be compared.
Preoperative and postoperative INCONTINENCE IMPACT QUESTIONNAIRE | 1 year
  Scores ranges from 0 to 21 AND a higher score indicates more severe symptoms and lower quality of life. Pre and postoperative values will be compared.

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziosmanpasa Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes